CLINICAL TRIAL: NCT04811443
Title: DEFENDOR: A Multicenter Prospective Observational Post-registration stuDy of Extimia® (INN: empEgfilrastim) to Evaluate Efficacy and saFEty in patieNts With soliD tumORs
Acronym: DEFENDOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Other Study IDs: BCD-017-01-NIS
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Patients With Solid Tumours Who Receive Myelosupressive Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with solid tumors who have received myelosupressive therapy
  Interventions: Drug: Empegfilgrastim

INTERVENTIONS:
Drug: Empegfilgrastim — Extimia®

SUMMARY:
This study was designed to evaluate the efficacy and safety of Extimia® (INN - empegfilgrastim) in reducing the frequency, duration of neutropenia, the incidence of febrile neutropenia and infections caused by febrile neutropenia in patients with solid tumours receiving myelosuppressive therapy

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Histologically verified diagnosis;
3. Age between 18 and 80 years;
4. If the patient had previously received chemotherapy for these indications, then it should be completed at least 30 days before the first administration of the study drug;
5. ECOG performance 0-2;
6. Haematology:

   * ANC ≥ 1,5 х 10(9) /L;
   * Platelets ≥ 100 х 10(9) /L;
   * Hemoglobin ≥ 90 g/L;
7. Biochemistry:

   * Creatinine ≤ 1,5 ULN;
   * Total bilirubin ≤ 1,5 ULN;
   * AST/ALT ≤ 2,5 ULN;
   * Alkaline phosphatase ≤ 5 ULN;
8. Life expectancy of at least 6 months from the date of the first drug administration in the study;
9. Ability of the patient to comply with the Protocol requirements.

Exclusion Criteria:

1. Documented hypersensitivity to empegfilgrastim, filgrastim, pegfilgrastim, and / or their constituent excipients: pegylated drugs, protein recombinant drugs;
2. Systemic use of antibiotics less than 72 hours before the first drug administration in the study;
3. Concurrent or less than 30 days before the start of the study, radiation therapy (with the exception of point radiation therapy for bone metastases); study;
4. Concurrent participation in clinical trials, participation in clinical trials within the previous 30 days, previous participation in this study;
5. Surgical treatment less than 21 days (3 weeks) prior to study enrollment; taking any experimental medications less than 30 days before enrollment in this study;
6. History of bone marrow or hematopoietic stem cell transplantation;
7. Presence of acute or active chronic infections;
8. Other diseases (with the exception of the main one) that could affect the assessment of the severity of the symptoms of the underlying disease: that may mask, enhance, change the symptoms of the underlying disease or cause clinical manifestations and changes in the data of laboratory and instrumental research methods;
9. Inability to administer the drug by intravenous infusion or subcutaneous injection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors who are prescribed myelosuppressive therapy with empegfilgrastim supportive therapy to reduce the frequency, duration of neutropenia, the incidence of febrile neutropenia (FN) and infections manifested by FN, as part of routine clinical practice according to the approved indications of the appropriate drugs.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-06-12 (Estimated); Study Completion 2022-06-12 (Estimated)

PRIMARY OUTCOMES:
Relative dose-intensity (RDI) of the myelosupressive therapy course | 12 months

SECONDARY OUTCOMES:
The incidence of febrile neutropenia with empegfilgrastim supportive therapy compared with historical control | 18 months
The incidence of neutropenia leading to a dose reduction of cytostatic drugs and / or an increase of the interval between cycles when using empegfilgrastim supportive therapy compared with historical controls | 18 months
RDI of chemotherapy courses performed in relation to nosology | 18 months
RDI of chemotherapy courses performed in relation to treatment regimen | 18 months
Any grade adverse events frequency | 18 months
Grade 3-4 adverse events frequency | 18 months
Serious adverse events frequency | 18 months
Frequency of study withdrawal due to adverse events | 18 months
The incidence of severe infections (grade 3-4) | 18 months
Frequency of antibiotic prescription | 18 months

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Regional Clinical Oncology Hospital, Yaroslavl, Yaroslavl Oblast
  - St. Josaphat Belgorod Regional Clinical Hospital, Belgorod
  - State Health Institution "Voronezh Region Clinical Oncology Dispansary", Voronezh

IPD SHARING:
Plan to Share IPD: No